CLINICAL TRIAL: NCT05959564
Title: A Chatbot Intervention for Reducing HPV Vaccine Hesitancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1960782-1
Record Dates: First submitted 2023-07-06; First posted 2023-07-25 (Actual); Results first posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-07

CONDITIONS: Cervical Cancer; Anal Cancer; Penile Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Anus Neoplasms; Penile Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Chatbot Condition (Experimental): After reading a standard CDC HPV vaccine message, participants will interact with a chatbot designed to deliver personalized HPV vaccine messages (i.e., tailored to their personalities).
  Interventions: Behavioral: Personalized Chatbot Intervention
- Non-Personalized Chatbot Condition (Experimental): After reading a standard CDC HPV vaccine message, participants will interact with a chatbot designed to deliver HPV vaccine messages, which are not tailored to their personalities.
  Interventions: Behavioral: Non-Personalized Chatbot Intervention
- No Chatbot Control Condition (Active Comparator): Participants will read a standard CDC HPV vaccine message without interacting with any chatbot that delivers additional messages.
  Interventions: Behavioral: No Chatbot Control

INTERVENTIONS:
Behavioral: Personalized Chatbot Intervention — In this intervention, participants will first see a standard CDC HPV vaccine message. After that they will be invited to interact with a chatbot designed to deliver additional HPV vaccine messages, which are tailored to their personalities.
  Arms: Personalized Chatbot Condition
Behavioral: Non-Personalized Chatbot Intervention — In this intervention, participants will first see a standard CDC HPV vaccine message. After that they will be invited to interact with a chatbot designed to deliver additional HPV vaccine messages, which are not tailored to their personalities.
  Arms: Non-Personalized Chatbot Condition
Behavioral: No Chatbot Control — In this intervention, participants will see a standard CDC HPV vaccine message only and will not interact with any chatbot.
  Arms: No Chatbot Control Condition

SUMMARY:
The goal of this project is to test the efficacy of a chatbot intervention for reducing HPV vaccine hesitancy among African American parents. An online experiment will be conducted to test the effectiveness of the chatbot intervention with African American parents. Results of this project will inform future communication interventions for reducing vaccine hesitancy among African American parents.

DETAILED DESCRIPTION:
The goal of this project is to test the efficacy of a chatbot intervention for reducing HPV vaccine hesitancy among African American parents. An online survey-experiment will be conducted. In the survey-experiment, participants will first answer questions related to their attitudes toward childhood vaccines and see a brief CDC message about HPV vaccine. Then they will be directed to interact with a chatbot designed to deliver personalized HPV vaccine messages (tailored to the participant's personality) or a similar chatbot with non-personalized messages. There will also be a control condition where participants will see the brief CDC message about HPV vaccine but will not interact with any chatbot. All participants will answer questions related to their attitudes toward HPV vaccination, intentions to vaccinate their children, as well as other message response measures.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Self-identify as Black or African American
* Parents of children under 18 years old
* Access to computer/laptop/mobile device and the Internet

Exclusion Criteria:

* Under 18 years
* Does not self-identify as Black or African American
* Not a parent of at least a child under 18 years old
* No access to computer/laptop/mobile device or the Internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 456 (Actual)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Nan, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park (Online Survey-Experiment), College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share anonymized data on data repositories such as the Open Science Framework.
Supporting Information: Study Protocol
Time Frame: After the study is published, for 5 years.
Access Criteria: All information is open to the public.

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Chatbot Condition: After reading a standard CDC HPV vaccine message, participants interacted with a chatbot designed to deliver personalized HPV vaccine messages (i.e., tailored to their personalities).
  Personalized Chatbot Intervention: In this intervention, participants first saw a standard CDC HPV vaccine message. After that they were invited to interact with a chatbot designed to deliver additional HPV vaccine messages, which were tailored to their personalities.
- Non-Personalized Chatbot Condition: After reading a standard CDC HPV vaccine message, participants interacted with a chatbot designed to deliver HPV vaccine messages, which were not tailored to their personalities.
  Non-Personalized Chatbot Intervention: In this intervention, participants first saw a standard CDC HPV vaccine message. After that they were invited to interact with a chatbot designed to deliver additional HPV vaccine messages, which were not tailored to their personalities.
- No Chatbot Control Condition: Participants read a standard CDC HPV vaccine message without interacting with any chatbot that delivers additional messages.
  No Chatbot Control: In this intervention, participants saw a standard CDC HPV vaccine message only and did not interact with any chatbot.
Period: Overall Study
Arm/Group | Personalized Chatbot Condition | Non-Personalized Chatbot Condition | No Chatbot Control Condition
Started | 152 | 154 | 150
Completed | 152 | 154 | 150
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Chatbot Condition | Non-Personalized Chatbot Condition | No Chatbot Control Condition | Total
Number analyzed (Participants) | 152 | 154 | 150 | 456
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.16 (10.55) | 37.80 (9.33) | 40.98 (10.77) | 39.96 (10.32)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 64 | 64 | 72 | 200
  Female | 87 | 87 | 77 | 251
  Non-binary | 1 | 3 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 152 | 154 | 150 | 456
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Education [Count of Participants; unit: Participants] — Education was measured by this question: What is the highest level of school you completed? The response categories included:
  Less than high school Some high school High school graduate Some college College graduate Post-college
  Participants
    Less than high school | 1 | 1 | 1 | 3
    Some high school | 0 | 2 | 1 | 3
    High school graduate | 14 | 12 | 13 | 39
    Some college | 49 | 49 | 33 | 131
    College graduate | 70 | 68 | 81 | 219
    Post-college | 18 | 22 | 21 | 61

OUTCOME MEASURES:

1. Primary Outcome: Attitudes Toward HPV Vaccination
Description: Participants' attitudes toward HPV vaccination were measured by seven questions such as "The HPV vaccine is beneficial for adolescents." The responses were recorded on 1 (strongly disagree) to 5 (strongly agree) scales. Final score was the average of all 7 questions.
Time Frame: baseline posttest (test took approximately 5 minutes to complete)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Chatbot Condition | Non-Personalized Chatbot Condition | No Chatbot Control Condition
Number analyzed (Participants) | 152 | 154 | 150
score on a scale | 3.86 (.84) | 3.96 (.86) | 3.41 (.85)

2. Primary Outcome: Intentions Toward HPV Vaccination
Description: Participants' intentions toward vaccinating their children against HPV were measured by three questions such as "I am likely to get my child/children the HPV vaccine." Responses were indicated on 1 (strongly disagree) to 5 (strongly agree) scales. The final score was the average of the three questions.
Time Frame: baseline posttest (test took approximately 5 minutes to complete)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Chatbot Condition | Non-Personalized Chatbot Condition | No Chatbot Control Condition
Number analyzed (Participants) | 152 | 154 | 150
score on a scale | 3.87 (1.17) | 3.95 (1.08) | 3.56 (1.18)

3. Secondary Outcome: Ratings of the Chatbot
Description: Ratings of the Chatbot were measured by nine questions such as "How would you describe the HPV chatbot you just interacted with? - Engaging" on 1 (strongly disagree) to 5 (strongly agree) scales. The final score was the average of the nine questions.
Time Frame: baseline posttest (test took approximately 5 minutes to complete)
Population: participants in the no chatbot control condition were not asked to rate the chatbot.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Chatbot Condition | Non-Personalized Chatbot Condition | No Chatbot Control Condition
Number analyzed (Participants) | 130 | 130 | 0
score on a scale | 4.10 (.79) | 4.16 (.70) |

ADVERSE EVENTS:
Description: Deaths and/or adverse events were not monitored/assessed as this was an online study where participants completed the survey on their own computer at a location of their choice.
Arm/Group | Personalized Chatbot Condition | Non-Personalized Chatbot Condition | No Chatbot Control Condition
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The online survey-experiment may not fully reflect how individuals typically encounter health messages in the real world. There is concern about ecology validity. Also the long-term effects of message exposure were not determined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT05959564/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT05959564/SAP_001.pdf
  • Informed Consent Form (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT05959564/ICF_002.pdf